CLINICAL TRIAL: NCT04577391
Title: Comparing the Effects of Modified Constraint-Induced Movement Therapy and Bimanual Training in Children With Hemiplegic Cerebral Palsy Mainstreamed in Regular School: A Randomized Controlled Study
Brief Title: Comparing the Effectiveness of mCIMT and Bimanual Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Hasan Bingöl, Academician (Lecturer, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 79236777-050.01.04
Record Dates: First submitted 2020-09-24; First posted 2020-10-06 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy
Keywords: upper limb; hand; bimanual training; constraint-induced movement therapy; ICF-CY; hemiplegic cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial: Work consisting of a clinical trial that involves at least one test treatment and one control treatment, concurrent enrollment and follow-up of the test- and control-treated groups, and in which the treatments to be administered are selected by a random process, such as the use of a random-numbers table
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes assessor was masked to group allocation/ participants were blinded to the presence of two different intervention approaches
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Constraint-Induced Movement Therapy (Experimental): Children's less affected hand was restricted through a mitt with a material sewn shut on the palmar face to promote the use of involved side as maximum as possible. Besides, if the participant attempted to use his/her less affected hand as an assistive, a bandage was also used to strap less affected upper limb to the trunk. Specific activities were selected according to deficit of interest, participant preference (on the condition of having potential effects on hand skills) and parent/guardian, or their teacher's request (e.g., drawing, painting, and eating). In case of activities requiring both hand use, such as stabilizing paper during the painting or holding the bricks of lego on the ground, the treating physiotherapist undertook the role of the child's dominant hand.
  Interventions: Other: Modified Constraint-Induced Movement Therapy
- Bimanual training (Active Comparator): BIT was administrated without any restrictive material on the non-involved upper limb, but instead, children were engaged in age-appropriate gross and fine motor bimanual activities. All targeted deficits of interest were addressed within the context of the selected activity.
  Interventions: Other: Bimanual Training

INTERVENTIONS:
Other: Modified Constraint-Induced Movement Therapy — Children's less affected hand was restricted through a mitt with a material sewn shut on the palmar face to promote the involved side's use, and unimanual gross and fine motor activities were practiced with the more affected hand. Besides, if the participant attempted to use his/her less affected hand as an assistive, a bandage was also used to strap less affected upper limb to the trunk. Specific activities were selected according to the deficit of interest, participant preference (on the condition of having potential effects on hand skills) and parent/guardian, or their teacher's request (e.g., drawing, painting, and eating).
  Arms: Modified Constraint-Induced Movement Therapy
Other: Bimanual Training — BIT was administrated without any restrictive material on the non-involved upper limb, but instead, children were engaged in age-appropriate gross and fine motor bimanual activities. All targeted deficits of interest were addressed within the context of the selected activity.
  Arms: Bimanual training

SUMMARY:
This study aimed to compare the effects of Modified Constraint-Induced Movement Therapy (mCIMT) and Bimanual Training (BIT) based on the International Classification of Functioning, Disability, and Health, Children &Youth (ICF-CY) conceptual framework. Our assumptions were that (1) mCIMT is more effective on outcomes representing all subdomains of ICF and (2) the possible improvements in the body structure and function, activity, and participation subdomains of ICF are intimately related to each other.

DETAILED DESCRIPTION:
Thirty-two children with spastic hemiplegic cerebral palsy (mean age 10.43 years [SD 2.9 years]; 15 females, 17 males) whose functional profiles associated with Manual Ability Classification System, Gross Motor Function Classification System, and Communication Function Classification System changed between level I-III were randomly distributed to one of the mCIMT or BIT groups with equivalent dosing frequency and intensity (10 weeks/3 days per week/2.5 hours per day). Outcome measures categorized according to the domains of International Classification of Functioning, Disability, and Health, Children &Youth (ICF-CY) framework were used to document body functions, activity, and participation outcomes. Assessments were carried out before (T1) and after treatment (T2), and at 16 weeks post-intervention (T3) by a physical therapist blinded to group allocation. Before the study entry, informed consent was obtained from the parents. General and specific contents related to each intervention were delivered as individual sessions at the school (one session per week) or group sessions with two participants at rehabilitation centers (two sessions per week).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of spastic hemiplegic cerebral palsy
* Must be able to attend primary or secondary school

Exclusion Criteria:

* Family-dependent problems interfering with participation in study sessions
* The presence of behavioral problems interfering with the assessment periods or intervention sessions

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in unimanual capacity on Upper Extremity Skills Test (QUEST) at 16 weeks | Baseline and week 16
  The Upper Extremity Skills Test (QUEST) is a criterion-referenced measurement tool, developed to evaluate upper extremity quality of movement in children with cerebral palsy.The Upper Extremity Skills Test has been validated for children with cerebral palsy aged 18 months to 12 years. Intra-rater reliability of the QUEST has been indicated to strong (ICC=0.96) in children with cerebral palsy aged eight and over.
Change from baseline in manual ability on ABILHAND-Kids at 16 weeks | Baseline and week 16
  ABILHAND-Kids is developed for children with cerebral palsy and measures a child's ability to manage 21 daily activities that require the use of the upper limbs. It measures the children's typical performance in daily life. ABILHAND-Kids is useful in reporting the functional performance of children with one affected side in the perspective of manual ability and has excellent test-retest reliability for Turkish children with cerebral palsy (ICC=0. 0.98)

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Bingöl, MSc, Principal Investigator — Muş Alparslan University
Locations (1):
- Mus Alparslan University, Muş, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fedrizzi E, Rosa-Rizzotto M, Turconi AC, Pagliano E, Fazzi E, Pozza LV, Facchin P; GIPCI Study Group. Unimanual and bimanual intensive training in children with hemiplegic cerebral palsy and persistence in time of hand function improvement: 6-month follow-up results of a multisite clinical trial. J Child Neurol. 2013 Feb;28(2):161-75. doi: 10.1177/0883073812443004. Epub 2012 May 10. PMID 22580904
- [Result] Gelkop N, Burshtein DG, Lahav A, Brezner A, Al-Oraibi S, Ferre CL, Gordon AM. Efficacy of constraint-induced movement therapy and bimanual training in children with hemiplegic cerebral palsy in an educational setting. Phys Occup Ther Pediatr. 2015 Feb;35(1):24-39. doi: 10.3109/01942638.2014.925027. Epub 2014 Jul 1. PMID 24983295
- [Result] Sakzewski L, Ziviani J, Boyd RN. Best responders after intensive upper-limb training for children with unilateral cerebral palsy. Arch Phys Med Rehabil. 2011 Apr;92(4):578-84. doi: 10.1016/j.apmr.2010.12.003. PMID 21440702
- [Result] Thompson AM, Chow S, Vey C, Lloyd M. Constraint-induced movement therapy in children aged 5 to 9 years with cerebral palsy: a day camp model. Pediatr Phys Ther. 2015 Spring;27(1):72-80. doi: 10.1097/PEP.0000000000000111. PMID 25521268
- [Derived] Bingol H, Gunel MK. Comparing the effects of modified constraint-induced movement therapy and bimanual training in children with hemiplegic cerebral palsy mainstreamed in regular school: A randomized controlled study. Arch Pediatr. 2022 Feb;29(2):105-115. doi: 10.1016/j.arcped.2021.11.017. Epub 2022 Jan 14. PMID 35039189